CLINICAL TRIAL: NCT03713567
Title: Clinical, Immunological and Microbiological Evaluation of Experimental Gingivitis and Peri-implant Mucositis in Patients With History of Agressive Periodontal Disease
Brief Title: Clinical, Immunological and Microbiological Evaluation of Experimental Gingivitis and Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Full Professor, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U1111-1217-5513
Record Dates: First submitted 2018-10-09; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Gingivitis; Mucositis
Keywords: Aggressive Periodontitis; Biomarkers; Microbiota; Dental Implants
MeSH Terms: conditions — Gingivitis; Mucositis; Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimentally induced plaque (Placebo Comparator): Induced inflammation by suspension of oral hygiene
  Interventions: Behavioral: Experimentally induced plaque
- Experimentally induced plaque GAP (Experimental): Induced inflammation by suspension of oral hygiene in patients with history of Generalized Aggressive periodontitis
  Interventions: Behavioral: Experimentally induced plaque

INTERVENTIONS:
Behavioral: Experimentally induced plaque — Experimentally induced plaque by suspension of oral hygiene only in the tested areas (tooth / implant), protected by a personalized stent made of plastic, according to the experimental gingivitis and mucositis model of 21 days of duration

SUMMARY:
The objective of this study is to evaluate, through clinical, microbiological and immunological tests, the changes during the experimental gingivitis and mucositis model, between teeth and implants, and between patients with a history of aggressive periodontitis and healthy individuals.

DETAILED DESCRIPTION:
The objective of this study is to evaluate, through clinical, microbiological and immunological tests, the changes during the experimental gingivitis and mucositis model, between teeth and implants, and between patients with a history of aggressive periodontitis and healthy individuals. 20 patients will be include, 10 healthy and 10 with a history of aggressive periodontitis. All patients must present the same type of implant and abutments, with prostheses in function for more than 6 months. They should also have a tooth located in the contralateral hemi-arch in a similar position, allowing a comparison with the implant. They will be submitted to the plaque-induced inflammation by suspension of oral hygiene only in the tested areas (tooth / implant), protected by a personalized stent made of plastic, according to the experimental gingivitis and mucositis model of 21 days of duration.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years,
* History of aggressive periodontitis diagnosed according to the Armitage classification (1999) and verified by the dental chart and time of radiographic bone emission, being in periodontal maintenance for a little more than 6 months (Test group).
* Presence of teeth and implants (unitary prostheses) in the mouth; in a similar and counter-lateral position in the arch. The implants are the same system, including protective and dimensions.
* Probing Depth <5mm, in the interest sites.
* Plaque Index ≤ 20% (Silness & Löe, 1964),
* Healthy patients
* Signature of free and informed consent.

Exclusion Criteria:

* Probing Depth> 5mm, in the interest sites.
* History of bone loss by peri-implantitis in the implant test.
* Smoking;
* Pregnancy;
* Presence of systemic disorders (diabetes, hypertension, heart disease or any other condition that could contraindicate periodontal surgery);
* Use of medications (immunosuppressants, phenytoin or anything else that might affect mucosal healing and repair);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Changes of Modified Gingival Index in five different periods | Baseline, 7 days, 14 days, 21 days, 42 days
  According to the method of Löe & Silness (1963) without the bleeding in the component of prueba.Measure at each visit 0 - absence of inflammation;
  1. - Light inflammation - slight color change and little alteration in gingival texture;
  2. - Moderate inflammation - moderate texture change, redness, edema, hypertrophy.
  3. - Severe inflammation - redness, hypertrophy.

SECONDARY OUTCOMES:
Changes of Angulated Bleeding Index in five different periods | Baseline, 7 days, 14 days, 21 days, 42 days
  0 - No bleeding.
  1. - Bleeding after probe stimulation.
  2. - Spontaneous bleeding
Changes of Plaque Index in five different periods | Baseline, 7 days, 14 days, 21 days, 42 days
  0 - Absence of plaque
  1. - A thin layer of plaque adhered to the free gingival margin and adjacent to the dental surface. The plaque can be seen in situ only after the use of an evidentiary solution or through the passage of the periodontal probe through the dental surface.
  2. - Moderate accumulation in the periodontal pocket, dental surface or gingival margin, seen with the naked eye.
  3. - Abundance of plaque in the periodontal pocket and / or on the dental surface and gingival margin.

OTHER OUTCOMES:
Changes of Gingival fluid in five different periods | Baseline, 7 days, 14 days, 21 days, 42 days
  Gingival fluid is collected from the fluid site and the paper strip is transfer to a Periotron 6000® (Pro Flow™, Amityville, NY, USA) for assessment of the fluid volume.

CONTACTS AND LOCATIONS:
Overall Officials: Tamires P Dutra, G, Principal Investigator — School of Odontology of Piracicaba - Unicamp
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Dutra TP, Freitas Monteiro M, Franca-Grohmann IL, Casarin RCV, Casati MZ, Silverio Ruiz KG, Kumar PS, Sallum EA. Clinical, immunological and microbiological evaluation of experimental peri-implant mucositis and gingivitis in subjects with Grade C, stage III/IV periodontitis background. J Clin Periodontol. 2024 Feb;51(2):209-221. doi: 10.1111/jcpe.13896. Epub 2023 Nov 8. PMID 37941050